CLINICAL TRIAL: NCT00165152
Title: A Randomized Study of Counseling Interventions for BRCA 1/2 Cancer Susceptibility Testing
Brief Title: Counseling Interventions for BRCA 1/2 Cancer Susceptibility Testing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Massachusetts General Hospital (Other); Beth Israel Deaconess Medical Center (Other); Medical University of South Carolina (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Judy E. Garber, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 98-120
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2012-08-09 (Estimated); Status verified 2012-08

CONDITIONS: Breast Cancer; Ovarian Cancer
Keywords: Genetic testing; BRCA1 gene; BRCA2 gene; Counseling interventions; Genetic counseling
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms; Fanconi Anemia, Complementation Group D1 | interventions — Genetic Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Genetic Counseling (Active Comparator)
  Interventions: Procedure: Genetic Counseling
- Informed Consent Counseling (Active Comparator)
  Interventions: Procedure: Informed Consent Counseling

INTERVENTIONS:
Procedure: Genetic Counseling — Two visits with a specially trained genetic counselor or nurse in conjunction with a medical oncologist and/or a medical specialist will be done in which information will be given either about genetic counseling or enhanced informed consent. These visits will be audio-taped to monitor how the project staff is covering the important information about testing.
  Arms: Genetic Counseling
Procedure: Informed Consent Counseling — Two visits with a specially trained genetic counselor or nurse in conjunction with a medical oncologist and/or a medical specialist will be done in which information will be given either about genetic counseling or enhanced informed consent. These visits will be audio-taped to monitor how the project staff is covering the important information about testing.
  Arms: Informed Consent Counseling

SUMMARY:
To evaluate two different ways of providing information about genetic testing for BRCA1 and BRCA2 alterations. The two forms of counseling are genetic counseling and enhanced informed consent which cover similar material but are organized differently.

DETAILED DESCRIPTION:
* Patients will have a blood sample drawn that will be analyzed for altered BRCA1 or BRCA2 genes. An alteration of BRCA1 or BRCA2 gene means there is an increased risk of developing breast and ovarian cancer.
* Patients participating in this study have either: 1) expressed an interest in testing for an underlying genetic factor that may account for the breast or ovarian cancer in their family; 2) have at least one relative that has been found to have a BRCA1 or BRCA2 alteration; 3) have a personal or family history of breast or ovarian cancer that is suggestive of a BRCA1 and BRCA2 alteration; or 4) has breast or ovarian cancer, or has at least one close relative with a history of breast or ovarian cancer and are a member of an ethnic group with increased frequency of BRCA1 and BRCA2 alterations.
* Patients will be randomized into one of two counseling groups. Two visits with a specially trained genetic counselor or nurse in conjunction with a medical oncologist and/or a medical specialist will be done in which information will be given either about genetic counseling or enhanced informed consent. These visits will be audio-taped to monitor how the project staff is covering the important information about testing.
* Throughout this study patients will be asked to complete questionnaires and psychological measures. These forms will be completed before and after the first visit, and a subset of them again at 2-4 weeks after the second visit, and at 4, 6, and 12 months.
* In addition 30 women will be asked to complete a 20-30 minute telephone interview with the program psychologist.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Member of a family in which a BRCA1 or BRCA2 deleterious germline mutation has been identified, whether or not the individual has had cancer herself; written documentation of the family mutation must be available for laboratory purposes during the testing process.
* Personal and/or family history of breast/ovarian/other cancer consistent with BRCA 1/2 heredity with posterior probability of carrying an altered gene
* Documentation of key family member cancer diagnoses is required

Exclusion Criteria:

* Males, will be offered BRCA 1/2 testing through other protocols
* Individuals unable to speak or write English
* Already participated in a genetic counseling program for BRCA1 or BRCA2 testing
* Life expectancy of less than 12 months.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 1998-07; Primary Completion 2001-09 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
To determine if genetic counseling yields better psycho-social and medical care utilization outcomes, compared to a medical model of informed consent for genetic testing. | 5 years

SECONDARY OUTCOMES:
To compare the financial costs incurred in the implementation of the two models and examine the utilization of medical and mental health services by participants in each condition during the follow-up period. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Judy Garber, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts